CLINICAL TRIAL: NCT03134118
Title: Single-arm, Multicentre, Phase II Study of Immunotherapy in Patients With Type B3 Thymoma and Thymic Carcinoma Previously Treated With Chemotherapy
Brief Title: Nivolumab in Patients With Type B3 Thymoma and Thymic Carcinoma (NIVOTHYM)
Acronym: NIVOTHYM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1525; 2015-005504-28 (EudraCT Number); ETOP 11-16 (Other: ETOP)
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Thymoma Type B3; Thymic Carcinoma
Keywords: Thymoma; Phase II; nivolumab; Thymic carcinoma
MeSH Terms: conditions — Thymoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Patients will be centrally registered and will receive nivolumab 240 mg IV every 2 weeks
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Patients will be centrally registered and will receive nivolumab 240 mg IV every 2 weeks
  Other Names: BMS-936558-01

SUMMARY:
The aim of the phase II Nivothym study is to collect data on activity and toxicity of nivolumab therapy in patients with thymic carcinoma or type B3 thymoma that previously received a first platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Relapsed/advanced thymoma B3 and thymic carcinoma not amenable to curative-intent radical treatment;

At least one previous line of platinum-based chemotherapy for advanced disease

* Patients treated with neo-adjuvant or adjuvant platinum based chemotherapy combined with radical surgical or as part of radical chemoradiotherapy are eligible if chemotherapy was completed less than 6 months before enrollment;
* Radiological progression documented per RECIST 1.1 during or after completion of previous line therapy;
* Presence of measurable disease according to RECIST 1.1.
* Disease status must be documented by full chest and upper abdomen (including adrenal glands) CT and/or MRI within 28 days of study enrollment. If clinically indicated, brain imaging must be performed
* At least 18 years;
* WHO Performance Status (PS) 0-2 Note: for the cohort of patient that will be treated with nivolumab and ipilimumab: PS 0-1
* Availability of FFPE tumor tissue (a tumour block or 10 unstained slides), notably for PD-L1 Immunohistochemistry (IHC) expression assessment. Archival material is allowed. Patients will be eligible to participate regardless of the level of PD-L1 expression, however tissue must be considered adequate (assessed by a local pathologist) for characterization of PD-L1 status as per procedure manual;
* Adequate hematological function:
* white blood count ≥ 2 × 109/L;
* haemoglobin >9 g/dL;
* platelet count >100 × 109/L;
* Adequate liver function:
* Total bilirubin <1.5 × ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL);
* ALT and/or AST <2.5 × ULN (< 4 x ULN in case of liver metastasis)
* alkaline phosphatase <5 × ULN;
* Adequate renal function: calculated creatinine clearance ≥50 mL/min (according to Cockroft- Gault, see below);
* Female CrCl = ((140 - age in years) x weight in kg x 0.85)/ 72 x serum creatinine in mg/dL;
* Male CrCl = ((140 - age in years) x weight in kg x 1.00)/72 x serum creatinine in mg/dL;
* Women of child bearing potential (WOCBP) must have a negative serum pregnancy test within 72 hours prior to the first dose of study treatment.

Note: women of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e. females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression or other reasons.

* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 5 months for a woman and 7 months for a man after the last study treatment. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Such methods include:
* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
* Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
* Intrauterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomized partner
* Sexual abstinence
* Female patients who are breast feeding should discontinue nursing prior to the first dose of study medication and must not be breast feeding during the trial treatment and for a period of at least 5 months following the last administration of trial drug(s).
* Before patient registration, written informed consent must be given according to ICH/GCP, and national/local regulations

Exclusion Criteria:

* No evidence of active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are clinically stable (i.e. without evidence of progression by imaging for at least four weeks prior to the enrollment and any neurologic symptoms have returned to baseline), and have not received steroids (for a total equivalent dose of more than 10mg of prednisone per day) for at least 7 days prior to enrollment;
* Prior treatment with anti-PD-1, anti-PD-L1/2, anti- CD137, CTLA-4 modulators;
* Current participation to any other clinical research nor treatment with an investigational agent or use of an investigational device within 4 weeks of the enrollment;
* Known history or current evidence of active Hepatitis B (e.g., HBsAg reactive) or C (e.g., HCV RNA[qualitative] is detected) or Human Immunodeficiency Virus (HIV) (HIV-1/2 antibodies);
* Known contra-indications for CT with IV contrast
* Chronic use of immunosuppressive agents and/or systemic corticosteroids or any use in the last 15 days prior to enrollment
* Corticosteroid use as premedication for IV contrast allergies/reactions is allowed;
* Daily prednisone at doses up to 10 mg or equivalent doses of any othe corticosteroid is allowed for example as replacement therapy
* No history of interstitial lung disease (ILD) OR pneumonitis (other than COPD exacerbation) that has required oral or IV steroids;
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (i.e., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed;
* Live vaccines within 30 days prior to the first dose of study therapy and while participating in study. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, H1N1 flu, rabies, BCG, and typhoid vaccine.
* Autoimmune paraneoplastic syndrome requiring immunosuppressive or dedicated treatment. A specific attention should be given in order to detect any minor myasthenia signs at enrollment; acetylcholine receptor antibodies will be systematically tested when symptoms are suggestive of a myasthenia;
* History of any other hematologic or primary solid tumor malignancy, unless in remission for at least 5 years. A pT1-2 prostatic cancer Gleason score < 6, superficial bladder cancer, non melanomatous skin cancer or carcinoma in situ of the cervix is eligible;
* Previous allogeneic tissue/solid organ transplant;
* Active infection requiring therapy;
* Surgery or chemotherapy related toxicity (toxicity resolved to grade 1, with the exception of alopecia, fatigue, neuropathy and lack of appetite /nausea);
* Severe comorbidities that in the opinion of the Investigator might hamper the participation to the study and/or the treatment administration;
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival Rate (PFSR) at month 6 | The Progression Free Survival Rate (PFSR) analysis will be performed at month 6

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 32 months after first patient in
Overall Survival (OS) | 32 months after first patient in
Toxicity according CTCAE version 4.03 | 32 months after first patient in
  This study will use the International Common Terminology Criteria for Adverse Events (CTCAE), version 4.03, for adverse event reporting.
Overall Response Rate (ORR) | 32 months after first patient in
  Overall Response Rate (ORR) will be measured according to RECIST 1.1
Disease Control Rate (DCR) | 32 months after first patient in
Duration of response | 32 months after first patient in

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Girard, Principal Investigator — Institut Curie, Paris, France; Solange Peters, Principal Investigator — University of Lausanne Hospitals
Locations (20):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen (UZA), Edegem
- France (8):
  - CHU de Brest, Brest
  - CHU de Lyon - Hopital Louis Pradel, Bron
  - Centre Francois Baclesse, Caen
  - CHU de Grenoble - La Tronche - Hôpital A. Michallon, La Tronche
  - Assistance Publique - Hopitaux de Marseille - Hopital Nord (APHM), Marseille
  - Institut Curie- Hopital de Paris, Paris
  - CHU Toulouse - Hopital Larrey, Toulouse
  - Gustave Roussy, Villejuif
- Netherlands (3):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Erasmus MC, Rotterdam
- Spain (2):
  - Vall d'Hebron Institut d'Oncologia, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
- UniversitaetsSpital Zurich, Zurich, Switzerland
- United Kingdom (4):
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre - Gartnavel General Hospital, Glasgow
  - Royal Marsden Hospital - Chelsea, London, London
  - Royal Marsden Hospital - Sutton, Surrey, Sutton
  - The Christie NHS Foundation Trust, Wythenshawe

REFERENCES:
- [Derived] Remon J, Girard N, Novello S, de Castro J, Bigay-Game L, Bernabe R, Greillier L, Mosquera J, Cousin S, Juan O, Sampayo M, Besse B. PECATI: A Multicentric, Open-Label, Single-Arm Phase II Study to Evaluate the Efficacy and Safety of Pembrolizumab and Lenvatinib in Pretreated B3-Thymoma and Thymic Carcinoma Patients. Clin Lung Cancer. 2022 May;23(3):e243-e246. doi: 10.1016/j.cllc.2021.07.008. Epub 2021 Jul 20. PMID 34393061